CLINICAL TRIAL: NCT04897945
Title: A Shared Decision Making Intervention for Diabetes Prevention in Women With a History of Gestational Diabetes Mellitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Intermountain Health Care, Inc. (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kenrik Duru, Professor Of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB#20-001558; R01DK127733 (NIH)
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-04

CONDITIONS: Gestational Diabetes Mellitus; Pre-diabetes; Diabetes Mellitus, Type 2
Keywords: Diabetes Prevention; Shared Decision Making
MeSH Terms: conditions — Diabetes, Gestational; Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shared decision-making with pharmacists (Experimental): Participants randomized to the intervention arm will have an in-person visit to complete the baseline survey, record the participant's weight and receive a pharmacist-coordinated shared decision making intervention. Intervention participants will have follow-up research assessments visits at 6, 12 and 24 months.
  Interventions: Behavioral: Shared decision-making for diabetes prevention
- Usual Care (No Intervention): Participants randomized to the usual care control arm will have an in-person visit with the research study team to complete the baseline survey and record the participant's weight. These participants will then return to usual care with research assessments at 6, 12 and 24 months follow-up.

INTERVENTIONS:
Behavioral: Shared decision-making for diabetes prevention — Pharmacists and/or nurses will engage patients with history of gestational diabetes mellitus using Healthwise (TM) Decision Tool to help match their personal preferences and values with treatment options, specifically lifestyle change will be referred to a CDC (Center for Disease Control and Prevention) recognized diabetes prevention program (DPP), and pharmacists will coordinate with primary care providers to prescribe metformin for patients interested in this treatment.
  Arms: Shared decision-making with pharmacists

SUMMARY:
Our goal is to test whether shared decision making for diabetes prevention can help women with a history of gestational diabetes mellitus (GDM) who are at high risk of developing type 2 diabetes (T2DM) increase weight loss and adoption of evidence based strategies to lower their risk of incident diabetes.

DETAILED DESCRIPTION:
Women with a history of gestational diabetes mellitus (GDM) are at high risk of developing type 2 diabetes (T2DM) but evidence from the Diabetes Prevention Program (DPP) indicates that lifestyle change and metformin use in this population are clinically equivalent, each reducing the incidence of T2DM by approximately 50%. Shared decision making (SDM) is an attractive approach in this situation where several options are available. We can use a decision aid to make the decision explicit, describe the available options with equipoise, elicit patient preferences, and help patients make an informed decision that is right for them. There are no existing studies evaluating SDM for diabetes prevention among women with a history of GDM. Therefore, this study aims to test the effectiveness of an RCT evaluating SDM for diabetes prevention on weight loss among overweight/obese women with a history of GDM and hemoglobin A1c between 5.7-6.4%, as well as uptake of lifestyle change and/or metformin use and other patient-reported outcomes (e.g., physical activity, eating patterns, patient activation, health-related quality of life). The study will recruit 310 patients from two large health care systems (n=155 from UCLA Health and n=155 from Intermountain Healthcare) who will be randomized to either usual care or in-person shared decision making for diabetes prevention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 54 (Adult)
* Females
* Most recent BMI ≥25 kg/m2 (or >23 if Asian American)
* History of gestational diabetes mellitus based on:
* Diagnostic code ICD10 or 1-hour glucose challenge test > 140 mg/dL, followed by 3-hour glucose tolerance test with TWO or more values. Cut-offs >= i. 95 at 0-hour ii. 180 at 1-hour iii. 155 at 2-hour iv. 140 at 3-hour
* History of prediabetes in prior 36 months defined by either

  1. most recent HbA1c 5.7-6.4% or
  2. most recent FPG 100-125 mg/dL or
  3. prior diabetes diagnostic codes + abnormal labs
* Patient at UCLA or Intermountain Healthcare Systems with provider visit or labs in prior 12 months

Exclusion Criteria:

* Delivery within the last 12 months at randomization
* History of diabetes (i.e., prior HbA1c 6.5% or above, or 2 or more fasting plasma glucose 125 or above, or prior diagnostic code)
* Any anti-glycemic medications or insulin use 12 months prior to randomization
* Most recent eGFR <45 ml/min
* BMI >60 kg/m2 at randomization
* History of any type of weight loss surgery 12 months prior to randomization
* Currently being treated for an eating disorder, such as anorexia or bulimia
* Currently pregnant or planning to get pregnant in the next 12 months
* Completed a prior prediabetes SDM consult anytime
* Currently enrolled OR have ever participated in any CDC certified Diabetes Prevention Program (DPP)
* Inability or concerns about doing >150 minutes of physical activity per week Currently taking a medication called metformin or have been prescribed metformin in the last 12-months
* History of metformin intolerance
* Unable to attend 3 virtual or in-person visits over the next 2 years at UCLA or Intermountain Healthcare
* Non-English primary language

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 310 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Weight change | 12 months
  Proportion with >5% weight loss

SECONDARY OUTCOMES:
Weight Change | 24 months
  Proportion with >5% weight loss
Uptake of DPP lifestyle program or metformin | 6 months
  1) Attending at least 9 of 16 of weekly lifestyle change sessions OR 2) Taking metformin (yes/no)
Health-related quality of life | 6, 12, and 24 months
  Short-form (SF-36) measure

CONTACTS AND LOCATIONS:
Overall Officials: Kenrik Duru, MD,MSHS, Principal Investigator — University of California, Los Angeles; Tannaz Moin, MD,MBA,MSHS, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Intermountain Healthcare System, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No